CLINICAL TRIAL: NCT06416085
Title: Psilocybin-assisted Existential, Attachment and RelationaL (PEARL) Therapy for Patients With Advanced Cancer: A Phase II Open-Label Trial
Brief Title: Psilocybin-assisted Existential, Attachment and RelationaL (PEARL) Therapy for Patients With Advanced Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PEARL; 21-5781 (Other: University Health Network)
Record Dates: First submitted 2024-01-14; First posted 2024-05-16 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Advanced Cancer; Stage IV Solid Tumor Cancer; Stage IV Sarcoma of Bone; Stage IV Lymphoma; Stage IV Melanoma; Endocrine Cancer
Keywords: Advanced Cancer
MeSH Terms: conditions — Osteosarcoma; Lymphoma; Melanoma; Endocrine Gland Neoplasms | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Psilocybin (Experimental)
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Single high-dose (25mg) capsule of psilocybin taken orally in the context of Psilocybin-assisted Existential, Attachment and RelationaL (PEARL) therapy

SUMMARY:
The PEARL Pilot is a phase II open-label trial. Participants will receive a single high-dose (25 mg) of psilocybin in the context of Psilocybin-assisted Existential, Attachment and RelationaL (PEARL) therapy.

DETAILED DESCRIPTION:
Individuals with advanced cancer often experience high levels of distress due to physical suffering, difficult treatment decisions, social isolation, and fear of death. While there are many treatment options for the management of physical symptoms associated with cancer, there are relatively few standard treatment approaches to help patients deal with psychological and existential suffering. Over the past decade, research has shown that psychotherapies incorporating existential, attachment and relational approaches can address the specific needs and challenges of the advanced cancer population and thus help to reduce distress. Simultaneously, recent research has shown that psilocybin-assisted psychotherapy, in which, an individual ingests the psychoactive drug within the carefully monitored therapeutic setting, can reduce end-of-life distress and greatly benefit those with advanced disease. The multidisciplinary team has combined these two evidence-based approaches into what the team calls Psilocybin-assisted Existential, Attachment and RelationaL (PEARL) therapy. PEARL therapy combines elements from psilocybin-assisted psychotherapy, including preparatory therapy sessions, a high-dose drug session, and integration sessions, with important elements from manualized individual psychotherapies designed for patients with advanced cancer. This study will assess the feasibility, acceptability, and safety of PEARL therapy among patients with advanced cancer. This study will yield important information about the feasibility of this type of therapy and contribute to the growing research around the efficacy of psychedelic-assisted therapies. This type of therapy has the potential to improve quality of life among those with advanced disease and careful research is needed to build upon previous findings to outline the necessary components of therapy and guide public policy, legislation, and clinical guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years of age.
2. Ability to speak and read English (patient to provide written informed consent and participate in PEARL intervention, as determined by study personnel).
3. Resident of Ontario.
4. No cognitive impairment indicated in medical record or by attending oncologist or palliative care physician.
5. Confirmed diagnosis of stage IV solid tumour cancers, sarcoma, endocrine, melanoma cancers, or stage 4 lymphoma with expected survival of greater than 6 months as determined by their oncologist or palliative care physician.
6. At least mild depressive symptoms, defined as >8 on the Patient Health Questionnaire-9 (PHQ-9) (Kroenke et la., 2001).
7. Interest in and ability to participate in and complete the PEARL intervention and protocol as outlined.
8. Participants who are sexually active and could become pregnant must be using effective birth control (per their physician), prior to study entry, during study participation, and for the duration of the study. Participants who are sexually active and could inseminate a partner must agree to use effective birth control after psilocybin administration until the end of study. For participants of child-bearing potential, a negative serum pregnancy test result is required at screening. A urine pregnancy test will be administered on the morning of psilocybin administration for applicable participants. Participants cannot be pregnant or nursing through the duration of the study.
9. If using prescribed medications or other substances, participants must agree to refrain from taking them if instructed by study investigators. These include:

   * not using any non-prescription medication, nutritional supplement, or herbal supplement except when approved by the treatment team (exceptions will be evaluated by the Investigator and will include acetaminophen, non-steroidal anti-inflammatory drugs, and common doses of vitamins and minerals),
   * not using nicotine for at least 2 hours before psilocybin administration, and not again until approximately 7 hours after psilocybin administration,
   * consuming approximately the same amount of caffeine-containing beverages (e.g., coffee, tea) that they consume on a usual morning before arriving at the treatment centre for the psilocybin session day,
   * not taking any as needed medications on the mornings of psilocybin sessions (with the exception of daily and as needed opioid pain medication),
   * refraining from using any psychoactive drugs, including alcoholic beverages, within 24 hours of the psilocybin administration.
10. Participants must have someone drive them after the session to where they are staying (home, hotel or another location), because psilocybin may affect their alertness and concentration on the evening of the dosing session.

Exclusion Criteria:

1. Primary cancer of the brain, or metastasis to the brain associated with clinically significant symptoms (e.g., affective, cognitive, personality-related, psychotic, or other symptoms, including seizures).
2. Symptoms consistent with delirium, psychosis, or other symptoms judged to be incompatible with establishment of rapport or safe exposure to psilocybin.
3. A history of past intolerability of psilocybin or other psychedelics.
4. Past/present psychiatric diagnoses including bipolar disorder, psychotic disorders, active substance use disorders or suicidality (as distinguished from desire for hastened death or readiness for death, per the discretion of the study team).
5. If participant is under 30 years of age and has first degree relative with a primary psychotic disorder.
6. Severe hypertension (defined as systolic blood pressure >150/or diastolic pressure >95) based on two readings on the same day. If the second reading remains over 150/95, the patient can be brought in for another reading on a different day. Patients can be re-screened for participation once blood pressure is adequately controlled.
7. Moderate or severe hepatic impairment, as defined by Child-Pugh class B or C, or elevations in AST or ALT greater than 3 times the upper limit of normal.
8. Severe renal impairment (defined as eGFR < 30).
9. Known paraneoplastic syndrome or "ectopic" hormone production by the primary tumor if incompatible with psilocybin, determined in consultation with the study palliative care physician. Patients could be enrolled if it is determined that the patient's condition is compatible with psilocybin administration.
10. Cardiovascular conditions including uncontrolled hypertension, angina, a clinically significant ECG abnormality (e.g., atrial fibrillation without rate control), transient ischemic attack in the last six months, stroke, peripheral or pulmonary vascular disease (no active claudication).
11. Uncontrolled epilepsy or history of seizures in past 6 months.
12. Participants with diabetes who are unable to skip a meal (lunch), or whose diabetes requires administration of medication more than twice daily, or who have had symptomatic hypoglycemia within the prior 30 days.
13. GI bleed in last 6 months.
14. Use of other agents that would be inappropriate to take with psilocybin in the judgement of the investigator. These agents may include psychoactive prescription medications (e.g., benzodiazepines, lithium, Selective serotonin reuptake inhibitors), medications having a primary pharmacological effect on serotonin-2a (5-HT2A) receptors (e.g., olanzapine), or medications that are monoamine oxidase (MAO) inhibitors, any potent metabolic inducers (e.g. rifamycin, rifampin, rifabutin, rifapentine, carbamazepine, phenytoin, phenobarbital, nevirapine, efavirenz, taxol, dexamethasone, St John's wort) or inhibitors (e.g. HIV protease inhibitors, itraconazole, ketoconazole, erythromycin, clarithromycin, troleandomycin).

Of note, in suitable patients, these medications may be paused or tapered between study enrolment and prior to the start of the intervention when it is deemed safe to do so. A safe and appropriate tapering regimen will then be developed based on the particular medication, on a case-by-case basis. If taking an MAO inhibitor, the psilocybin session will not be conducted until at least 5 half-lives of the agent have elapsed after the last dose. Patients prescribed opioids will be allowed to take their usual dose regimen for analgesia, including the use of as needed analgesic medications on psilocybin session days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Recruitment feasibility as assessed by the number of patients who consent/number of patients who meet eligibility criteria. | 24 months
  Used to assess feasibility of PEARL therapy.
Retention feasibility as assessed by the number of patients completing primary endpoint measures/number of patients consented. | 24 months
  Used to assess feasibility of PEARL therapy.
Adherence feasibility as assessed by the number of patients completing all PEARL sessions/number of patients consented. | 24 months
  Used to assess feasibility of PEARL therapy.
Acceptability of PEARL therapy from the perspective of advanced cancer patients obtained through qualitative interviews. | 24 months
  Participants will be interviewed regarding their experiences with PEARL, including acceptability and perceived positive and negative effects of the intervention, with a semi-structured interview guide.
Safety of PEARL therapy. | 24 months
  Safety will be assessed throughout the trial. Adverse events (AEs) attributed to psilocybin will be monitored for and recorded after the psilocybin session. This study will use CTCAE v5.0 to assess AEs.
  Serious adverse events (SAEs) will be tracked until study completion and will be defined as any adverse drug experience that: results in death; that is life-threatening (i.e. any AE that places the participant, in the view of the investigators, at immediate risk of death from the reaction as it occurs); requires hospital admission; results in persistent or significant disability (i.e. a substantial disruption of a person's ability to conduct normal life functions); or may jeopardize the participant or necessitate medical intervention to prevent one of the aforementioned criteria.

SECONDARY OUTCOMES:
Patient perspectives on the clinical relevance of potential PEARL therapy outcomes: Death anxiety in advanced cancer patients as assessed with the DADDS. | 24 months
  The Death and Dying Distress Scale (DADDS) is a 15-item self-report measure designed for populations facing imminent death and addresses fears about the dying process, and about lost opportunities and self-perceived burden placed on others as a result of impending mortality. Total score range is 0 to 75. Higher scores indicate greater death-related distress.
Patient perspectives on the clinical relevance of potential PEARL therapy outcomes: Depressive symptoms as assessed with the PHQ-9. | 24 months
  The Patient Health Questionnaire-9 (PHQ-9) is a 9-item self-report scale measuring depressive symptoms. Total score range is 0 to 27. Higher scores indicate greater severity of depression.
Patient perspectives on the clinical relevance of potential PEARL therapy outcomes: Anxiety symptoms as assessed with the GAD-7. | 24 months
  The Generalized Anxiety Disorder-7 (GAD-7) is a 7-item self-report scale used to screen for and measure anxiety symptoms. Total score range is 0 to 21. Higher scores indicate higher levels of anxiety.
Patient perspectives on the clinical relevance of potential PEARL therapy outcomes: Loss of meaning and purpose, disheartenment and helplessness as assessed with the DS. | 24 months
  The Demoralization Symptoms (DS) is a 24-item self-report measure that assesses loss of meaning and purpose, disheartenment, and helplessness. Total score range is 0 to 96. Higher scores indicate higher levels of demoralization.
Patient perspectives on the clinical relevance of potential PEARL therapy outcomes: Overall measure of spiritual well-being, meaning/peace and faith as assessed with the FACIT-Sp. | 24 months
  The Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being (FACIT-Sp) is a 12-item scale designed to measure important aspects of spirituality including sense of meaning in one's life, harmony, peacefulness and a sense of comfort and strength from one's faith. Total score range is 0 to 48. Higher scores indicate higher spiritual well-being.
Patient perspectives on the clinical relevance of potential PEARL therapy outcomes: Broad quality of life construct in patients facing end of life as assessed with the QUAL-EC. | 24 months
  The Quality of Life at the End of Life-Cancer (QUAL-EC) is a 17-item measure that includes subscales which assess symptom impact, preparation for end of life (i.e., the extent to which the family is prepared and financial plans have been made), relationship with healthcare providers (i.e., the extent to which patients feel informed and are able to participate in decisions about their care) and sense of life completion (i.e., being able to share important things and feel connected to others). For Symptom Control, score range is 3 to 15, with higher scores reflecting greater symptom control; for the Relationship with Healthcare Provider, score range is 5 to 25, with higher scores reflecting a better relationship with healthcare providers; for the Preparation for End-of-Life, score range is 4 to 20, with higher scores reflecting greater preparation for end-of-life; and the for Life Completion, score range is 5 to 25, with higher scores reflecting a greater sense of life completion.
Patient perspectives on the clinical relevance of potential PEARL therapy outcomes: Desire for death in the medically ill as assessed with the SAHD. | 24 months
  The Schedule of Attitudes Toward Hastened Death (SAHD) is a 20-item self-report measure of desire for death in the medically ill. Total score range is 0 to 20. Higher scores indicate greater desire for death.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Hales, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

REFERENCES:
- [Background] Albers G, Echteld MA, de Vet HC, Onwuteaka-Philipsen BD, van der Linden MH, Deliens L. Evaluation of quality-of-life measures for use in palliative care: a systematic review. Palliat Med. 2010 Jan;24(1):17-37. doi: 10.1177/0269216309346593. Epub 2009 Oct 20. PMID 19843620
- [Background] Breitbart W, Rosenfeld B, Gibson C, Pessin H, Poppito S, Nelson C, Tomarken A, Timm AK, Berg A, Jacobson C, Sorger B, Abbey J, Olden M. Meaning-centered group psychotherapy for patients with advanced cancer: a pilot randomized controlled trial. Psychooncology. 2010 Jan;19(1):21-8. doi: 10.1002/pon.1556. PMID 19274623
- [Background] Griffiths RR, Johnson MW, Carducci MA, Umbricht A, Richards WA, Richards BD, Cosimano MP, Klinedinst MA. Psilocybin produces substantial and sustained decreases in depression and anxiety in patients with life-threatening cancer: A randomized double-blind trial. J Psychopharmacol. 2016 Dec;30(12):1181-1197. doi: 10.1177/0269881116675513. PMID 27909165
- [Background] Grossman CH, Brooker J, Michael N, Kissane D. Death anxiety interventions in patients with advanced cancer: A systematic review. Palliat Med. 2018 Jan;32(1):172-184. doi: 10.1177/0269216317722123. Epub 2017 Aug 8. PMID 28786328
- [Background] Kissane DW, Wein S, Love A, Lee XQ, Kee PL, Clarke DM. The Demoralization Scale: a report of its development and preliminary validation. J Palliat Care. 2004 Winter;20(4):269-76. PMID 15690829
- [Background] Krause S, Rydall A, Hales S, Rodin G, Lo C. Initial validation of the Death and Dying Distress Scale for the assessment of death anxiety in patients with advanced cancer. J Pain Symptom Manage. 2015 Jan;49(1):126-34. doi: 10.1016/j.jpainsymman.2014.04.012. Epub 2014 May 28. PMID 24878066
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Lo C, Hales S, Zimmermann C, Gagliese L, Rydall A, Rodin G. Measuring death-related anxiety in advanced cancer: preliminary psychometrics of the Death and Dying Distress Scale. J Pediatr Hematol Oncol. 2011 Oct;33 Suppl 2:S140-5. doi: 10.1097/MPH.0b013e318230e1fd. PMID 21952572
- [Background] Morita T, Murata H, Kishi E, Miyashita M, Yamaguchi T, Uchitomi Y; Japanese Spiritual Care Task Force. Meaninglessness in terminally ill cancer patients: a randomized controlled study. J Pain Symptom Manage. 2009 Apr;37(4):649-58. doi: 10.1016/j.jpainsymman.2008.04.017. Epub 2008 Oct 1. PMID 18834700
- [Background] Rodin G, Lo C, Mikulincer M, Donner A, Gagliese L, Zimmermann C. Pathways to distress: the multiple determinants of depression, hopelessness, and the desire for hastened death in metastatic cancer patients. Soc Sci Med. 2009 Feb;68(3):562-9. doi: 10.1016/j.socscimed.2008.10.037. Epub 2008 Dec 7. PMID 19059687
- [Background] Rodin G, Lo C, Rydall A, Shnall J, Malfitano C, Chiu A, Panday T, Watt S, An E, Nissim R, Li M, Zimmermann C, Hales S. Managing Cancer and Living Meaningfully (CALM): A Randomized Controlled Trial of a Psychological Intervention for Patients With Advanced Cancer. J Clin Oncol. 2018 Aug 10;36(23):2422-2432. doi: 10.1200/JCO.2017.77.1097. Epub 2018 Jun 29. PMID 29958037
- [Background] Rosenfeld B, Breitbart W, Galietta M, Kaim M, Funesti-Esch J, Pessin H, Nelson CJ, Brescia R. The schedule of attitudes toward hastened death: Measuring desire for death in terminally ill cancer patients. Cancer. 2000 Jun 15;88(12):2868-75. doi: 10.1002/1097-0142(20000615)88:123.0.co;2-k. PMID 10870074
- [Background] Smith KA, Harvath TA, Goy ER, Ganzini L. Predictors of pursuit of physician-assisted death. J Pain Symptom Manage. 2015 Mar;49(3):555-61. doi: 10.1016/j.jpainsymman.2014.06.010. Epub 2014 Aug 10. PMID 25116913
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Steinhauser KE, Clipp EC, Bosworth HB, McNeilly M, Christakis NA, Voils CI, Tulsky JA. Measuring quality of life at the end of life: validation of the QUAL-E. Palliat Support Care. 2004 Mar;2(1):3-14. doi: 10.1017/s1478951504040027. PMID 16594230
- [Derived] Richardson C, Chan C, Macgregor E, Hare C, Hannon B, Black S, Schneider E, Buchman D, Wang S, Rac V, Abrahamyan L, Huszti E, Nissim R, Li M, Zimmermann C, Hapke E, Rosenbaum D, Hales S. Psilocybin-assisted Existential, Attachment and RelationaL (PEARL) therapy for patients with advanced cancer: protocol for a multi-method feasibility trial. Pilot Feasibility Stud. 2025 Oct 28;11(1):126. doi: 10.1186/s40814-025-01706-5. PMID 41152967